CLINICAL TRIAL: NCT04542057
Title: A Phase III Randomized, Double-Blind, Placebo-Controlled Study to Evaluate the Efficacy and Safety of Ensifentrine Over 24 Weeks in Patients With Moderate to Severe Chronic Obstructive Pulmonary Disease
Brief Title: A Phase 3 Trial to Evaluate the Safety and Efficacy of Ensifentrine in Patients With COPD
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Verona Pharma plc (Industry)
Collaborators: Iqvia Pty Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: RPL554-CO-302
Record Dates: First submitted 2020-09-01; First posted 2020-09-09 (Actual); Results first posted 2023-07-24 (Actual); Last update posted 2023-10-16 (Actual); Status verified 2023-10

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — ensifentrine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Arm 1 (Experimental): Ensifentrine Nebulized Suspension; 3 mg twice daily for 24 weeks
  Interventions: Drug: Ensifentrine
- Arm 2 (Placebo Comparator): Ensifentrine Placebo Nebulized Solution; twice daily for 24 weeks
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ensifentrine — Dosage Formulation:
  Ensifentrine Nebulizer suspension Dosage 3mg Frequency: Twice Daily for 24 weeks
  Arms: Arm 1
Drug: Placebo — Dosage Formulation:
  Ensifentrine Placebo Nebulizer solution Frequency: Twice Daily for 24 weeks
  Arms: Arm 2

SUMMARY:
The purpose of this study is to determine if ensifentrine is safe and effective for the treatment of patients with moderate to severe Chronic Obstructive Pulmonary Disease (COPD).

ELIGIBILITY:
Inclusion Criteria:

Informed Consent

1. Capable of giving informed consent indicating that they understand the purpose of the study and study procedures and agree to comply with the requirements and restrictions listed in the informed consent form (ICF).

   Age and Sex
2. Age: Patient must be 40 to 80 years of age inclusive, at the time of Screening.
3. Sex:

   * Males are eligible to participate if they agree to use contraception as described in the contraceptive guidance from Screening and throughout the study and for at least 30 days after the last dose of blinded study medication.
   * Females are eligible to participate if they are not pregnant, not breastfeeding, and at least one of the following conditions apply:

     1. Not a woman of childbearing potential (WOCBP). Or
     2. A WOCBP who agrees to follow the contraceptive guidance from Screening and throughout the study and for at least 30 days after the last dose of blinded study medication.

   Smoking History
4. Smoking History: Current or former cigarette smokers with a history of cigarette smoking ≥10 pack years at Screening (Visit 0) [number of pack years = (number of cigarettes per day / 20) × number of years smoked (eg, 20 cigarettes per day for 10 years, or 10 cigarettes per day for 20 years)]. Pipe and/or cigar use cannot be used to calculate pack-year history. Former smokers are defined as those who have stopped smoking for at least 6 months prior to Visit 0. Smoking cessation programs are permitted during the study.

   COPD Diagnosis, Symptoms, Severity and Maintenance Therapy
5. COPD Diagnosis: Patients with an established clinical history of COPD as defined by the American Thoracic Society (ATS)/European Respiratory Society (ERS) guidelines (Celli BR, 2004) with symptoms compatible with COPD.
6. COPD Symptoms: A score of ≥2 on the Modified Medical Research Council (mMRC) Dyspnea Scale.
7. COPD Severity:

   1. Pre- and Post-albuterol/salbutamol FEV1/FVC ratio of <0.70.
   2. Post-albuterol/salbutamol FEV1 ≥30 % and ≤70% of predicted normal calculated using the National Health and Nutrition Examination Survey III.
8. Maintenance Therapy: Patients on no maintenance/background therapy or patients on stable maintenance LAMA or LABA therapy are eligible. Patients taking maintenance LAMA or LABA therapy must demonstrate stable use of the maintenance LAMA or LABA therapy for at least 3 months prior to Screening and agree to continue use for the duration of the study. Background maintenance LAMA or LABA bronchodilator therapy will be capped at 50% of patients.

   Other Requirements for Inclusion
9. Capable of withholding SABAs for 4 hours prior to initiation of any spirometry. Patients in the maintenance LAMA or LABA therapy stratum must be capable of withholding Twice-Daily maintenance LAMA or LABA for 24 hours and Once-Daily maintenance LAMA or LABA for 48 hours prior to initiation of any spirometry.
10. Capable of using the study nebulizer correctly and complying with all study restrictions and procedures.
11. Ability to perform acceptable spirometry in accordance with ATS/ERS guidelines.

Randomization Criteria Criteria for Inclusion at Randomization

1. Symptoms of COPD: A score of ≥2 on the mMRC Dyspnea Scale.
2. Completion of the e-Diary at least 5 of the last 7 days of the Run-in period.

Exclusion Criteria:

Current Condition or Medical History

1. History of life-threatening COPD including Intensive Care Unit admission and/or requiring intubation.
2. Hospitalizations for COPD, pneumonia, or Corona Virus Disease 2019 (COVID-19) in the 12 weeks prior to Screening and/or a positive COVID-19 test result indicating an active infection at Screening. Patients with COVID-19 antibodies from a previous exposure with no active infection are not excluded.
3. COPD exacerbation requiring oral or parenteral steroids within 3 months of Screening.
4. Previous lung resection or lung reduction surgery within 1-year of Screening.
5. Long term oxygen use defined as oxygen therapy prescribed for greater than 12 hours per day. As needed oxygen use (≤12 hours per day) is not exclusionary.
6. Pulmonary rehabilitation, unless such treatment has been in a stable maintenance phase for 4 weeks prior to Visit 1 and remains stable during the study.
7. Lower respiratory tract infection within 6 weeks of Screening.
8. Other respiratory disorders including, but not limited to, a current diagnosis of asthma, active tuberculosis, lung cancer, sarcoidosis, lung fibrosis, interstitial lung diseases, unstable sleep apnea, known alpha-1 antitrypsin deficiency, core pulmonale, clinically significant pulmonary hypertension, clinically significant bronchiectasis, or other active pulmonary diseases.
9. Major surgery (requiring general anesthesia) in the 6 weeks prior to Screening, lack of full recovery from surgery at Screening, or planned surgery through the end of the study.
10. Historical or current evidence of clinically significant cardiovascular disease defined as any disease that in the opinion of the Investigator would put the safety of the patient at risk through participation or which could affect the efficacy or safety analysis if the disease/condition were to exacerbate during the study, including, but not limited to:

    * Myocardial infarction or unstable angina within 6 months prior to Screening.
    * Unstable or life-threatening cardiac arrhythmia requiring intervention within 3 months prior to Screening.
    * Diagnosis of New York Heart Association Class III and Class IV heart failure.
11. Chronic uncontrolled disease including, but not limited to, endocrine, active hyperthyroidism, neurological, hepatic, gastrointestinal, renal, hematological, urological, immunological, psychiatric, or ophthalmic diseases that the Investigator believes are clinically significant.
12. Unstable liver disease defined by the presence of ascites, encephalopathy, coagulopathy, hypoalbuminemia, esophageal or gastric varices or persistent jaundice, cirrhosis, known biliary abnormalities (except for Gilbert's syndrome or asymptomatic gallstones).
13. History of or current malignancy of any organ system, treated or untreated within the past 5 years, except for localized basal or squamous cell carcinoma of the skin.
14. Findings on physical examination that an investigator considers to be clinically significant at Screening.

    Prior/Concomitant Therapy
15. Use of prohibited medications within the time intervals

    History or Suspicion of Drug or Alcohol Abuse
16. Current or history of past drug or alcohol abuse within the past 5 years.

    Laboratory and Other Diagnostic Parameters
17. Glomerular Filtration Rate (eGFR) <30 mL/min. The Chronic Kidney Disease Epidemiology Collaboration Creatinine (2009) calculation will be used.
18. Alanine aminotransferase (ALT) ≥ 2 x upper limit of normal (ULN), alkaline phosphatase and/or bilirubin > 1.5 x ULN (isolated bilirubin >1.5 x ULN is acceptable if bilirubin is fractionated and direct bilirubin <35%).
19. Hepatitis B antibody:

    * Positive findings for both Hepatitis B surface antigen (HBsAg) and Hepatitis B core antibody (anti-HBc) are excluded, as this indicates acute or chronic infection.
    * Negative findings for HBsAg and Hepatitis B surface antibody (anti-HBs) but positive findings for anti-HBc are excluded as this may indicate current or resolving infection.
    * Positive findings for anti-HBc and anti-HBs but negative findings for HBsAg are not excluded, as this indicates immunity due to natural infection.
    * Positive findings for anti-HBs but negative findings for HBsAg and anti-HBc are not excluded, as this indicates immunity due to hepatitis B vaccination.
20. Hepatitis C antibody positive.
21. Any other abnormal hematology, biochemistry, or viral serology deemed by an investigator to be clinically significantly abnormal. Abnormal chemistry and/or hematology may be repeated during Screening.
22. Chest X-ray (CXR; posterior-anterior) at Screening, or in the 12 months prior to Screening with clinically significant abnormalities not attributable to COPD. If a CXR within the past 12 months is not available but a computerized tomography (CT) scan within the same time period is available, the CT scan may be reviewed in place of a CXR. For subjects in Germany, if a CXR or CT scan is not available in the 12 months prior to Screening, the subject is not eligible for the study.
23. Electrocardiogram (ECG) finding that is significantly abnormal on the 12-lead ECG obtained at Screening.

    Other Exclusions
24. Use of an experimental drug within 30 days or 5 half-lives of Screening, whichever is longer, and/or participation in a study treatment-free follow-up phase of a clinical trial within 30 days prior to Screening.
25. Use of an experimental medical device or participation in a follow-up phase of an experimental medical device clinical trial within 30 days prior to Screening.
26. Intolerance or hypersensitivity to albuterol/salbutamol or ensifentrine (RPL554) or any of its excipients/components.
27. Prior receipt of blinded study medication in an ensifentrine (RPL554) study.
28. Affiliation with the investigator site, including an Investigator, Sub-Investigator, study coordinator, study nurse, other employee of participating investigator or study site or a family member of the aforementioned.
29. Inability to read, understand, and/or complete questionnaires (in the opinion of the Investigator).
30. A disclosed history or one known to the Investigator of significant non-compliance in previous investigational studies or with prescribed medications.
31. Any other reason that the Investigator considers makes the patient unsuitable to participate.

Criteria for Exclusion from Randomization

1. COPD exacerbation or lower respiratory tract infection between Screening and Randomization (defined as use of any additional treatment other than current treatment and rescue medication and/or emergency department or hospital visit). Patients with a severe COPD exacerbation that requires hospitalization may not be rescreened.
2. Positive COVID-19 result at Screening or between Screening and Randomization.
3. Prohibited medication use between Screening Visit 0 and Visit 1.
4. Significantly abnormal ECG finding on the 12-lead ECG obtained at Screening as assessed by the investigator or site medical doctor/medically qualified person or on the pre-dose (prior to randomization) ECG obtained at Visit 1. In the event that the central ECG reviewer discovers a significant ECG abnormality on the Visit 1 ECG, the patient will be discontinued.
5. Did not meet one or more of the Inclusion Criteria or met one or more of the Exclusion Criteria.

Ages: 40 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 790 (Actual)
Dates: Start 2020-09-22 (Actual); Primary Completion 2022-05-03 (Actual); Study Completion 2022-07-06 (Actual)

CONTACTS AND LOCATIONS:
Locations (130):
- United States (77):
  - Wright Clinical Research, LLC, Alabaster, Alabama
  - SEC Clinical Research, Andalusia, Alabama
  - Jasper Summit Research LLC, Jasper, Alabama
  - Pulmonary Associates Clinical Trials, Phoenix, Arizona
  - Elite Clinical Studies LLC, Phoenix, Arizona
  - Clinical Research Institute of Arizona, LLC, Sun City West, Arizona
  - Premier Medical Group, Bakersfield, California
  - Antelope Valley Clinical Trials, Lancaster, California
  - Downtown LA Research Center, Inc., Los Angeles, California
  - UCLA Medical Center, Los Angeles, California
  - California Medical Research Associates, Northridge, California
  - Center for Clinical Trials of Sacramento, Inc., Sacramento, California
  - Integrated Research Center, San Diego, California
  - Institute of HealthCare Assessment, Inc., San Diego, California
  - Alpine Clinical Research Center, Boulder, Colorado
  - Innovative Research of West Florida, Clearwater, Florida
  - Clinical Research of West Florida, Inc., Clearwater, Florida
  - Accel Research Sites - DeLand Clinical Research Unit, DeLand, Florida
  - Riverside Clinical Research, Edgewater, Florida
  - Medical Research of Central Florida, Leesburg, Florida
  - Axcess Medical Research, Loxahatchee Groves, Florida
  - Research Institute of South Florida, Miami, Florida
  - Advanced Medical Research Institute, Miami, Florida
  - Clinical Trials of Florida. LLC, Miami, Florida
  - South Medical Research Group, Inc., Miami, Florida
  - ProCare Clinical Research, Miami Gardens, Florida
  - HMD Research, LLC, Orlando, Florida
  - Florida Institute for Clinical Research, Orlando, Florida
  - Sarasota Clinical Research, Sarasota, Florida
  - Coastal Pulmonary Critical Care, St. Petersburg, Florida
  - Pasadena Center for Medical Research, LLC, St. Petersburg, Florida
  - Clinical Research of West Florida, Inc., Tampa, Florida
  - Clinical Research Trials of Florida, Inc., Tampa, Florida
  - Florida Pulmonary Research Institute, LLC, Winter Park, Florida
  - AMR New Orleans, New Orleans, Louisiana
  - Genesis Clin RES& Consulting, Fall River, Massachusetts
  - Minnesota Lung Center, Edina, Minnesota
  - Minnesota Lung Center, Woodbury, Minnesota
  - Midwest Chest Consultants, Saint Charles, Missouri
  - Montana Medical Research Inc., Missoula, Montana
  - Mid Hudson Medical Research, New Windsor, New York
  - CHEAR Center LLC, The Bronx, New York
  - Carolina Clinical Research, Charlotte, North Carolina
  - American Health Research, Charlotte, North Carolina
  - Clinical Research of Gastonia, Gastonia, North Carolina
  - PharmQuest LLC, Greensboro, North Carolina
  - Monroe Biomedical Research, Monroe, North Carolina
  - Clinical Research of Lake Norman, Mooresville, North Carolina
  - Carolina Research Center, Inc., Shelby, North Carolina
  - Aventiv Research Inc., Columbus, Ohio
  - Remington Davis Clinical Research, Columbus, Ohio
  - Aventiv Research, Dublin, Ohio
  - OK Clinical Research, LLC, Edmond, Oklahoma
  - Velocity Clinical Research, Medford (Crisor, LLC), Medford, Oregon
  - Safe Harbor Clinical Research, East Providence, Rhode Island
  - VitaLink Research Anderson, Anderson, South Carolina
  - Lowcountry Lung and Critical Care, P.A., Charleston, South Carolina
  - VitaLink Research Columbia, Columbia, South Carolina
  - Piedmont Research Partners, Fort Mill, South Carolina
  - VitaLink Research Gaffney, Gaffney, South Carolina
  - VitaLink Research - Greenville, Greenville, South Carolina
  - Clinical Research of Rock Hill, Rock Hill, South Carolina
  - Spartanburg Medical Research, Spartanburg, South Carolina
  - VitaLink Research Spartanburg, Spartanburg, South Carolina
  - CU Pharmaceutical Research, Union, South Carolina
  - MultiSpecialty Clinical Research, Inc., Johnson City, Tennessee
  - New Phase Research Development, Knoxville, Tennessee
  - PnP Research, Amarillo, Texas
  - TTS Research, Boerne, Texas
  - Corsicana Medical Research, PLLC, Corsicana, Texas
  - Houston Pulmonary and Sleep Allergy and Asthma Associates, Cypress, Texas
  - Metroplex Pulmonary and Sleep Center, McKinney, Texas
  - Diagnostics Research Group, San Antonio, Texas
  - Element Research Group, San Antonio, Texas
  - Sherman Clinical Research, Sherman, Texas
  - DM Clinical Research, Tomball, Texas
  - Manassas Clinical Research Center, Manassas, Virginia
- Belgium (4):
  - UZA, Edegem
  - C.H.R. de la Citadelle, Liège
  - Private Practice RESPISOM Namur, Namur
  - AZ Delta, Roeselare
- Bulgaria (18):
  - MHAT 'Puls' AD, Blagoevgrad
  - Medical Centre "Asklepii", OOD, Dupnitsa
  - MHAT 'Dr. Stamen Iliev', AD, Montana
  - SHATPPD - Pazardzhik, EOOD, Pazardzhik
  - SHATPD Pernik, Pernik
  - Medical Center- Prolet Ltd, Rousse
  - SHATPPD-Ruse EOOD, Rousse
  - University First MHAT-Sofia, "St. Joan Krastitel" EAD, Sofia
  - Fifth MHAT - Sofia EAD, Sofia
  - NMTH "Tsar Boris III", Sofia
  - MHAT "Lyulin", EAD, Sofia
  - DCC "Alexandrovska", EOOD, Sofia
  - Diagnostic Consultation Center CONVEX EOOD, Sofia
  - Medical Center "Nov Rehabilitatsionen Tsentar", EOOD, Stara Zagora
  - Medical Center "ResearchExpert", OOD, Varna
  - MC "Tara", OOD, Veliko Tarnovo
  - SHATPPD "Dr. Treyman" EOOD, Veliko Tarnovo
  - SHATPPD - Vratsa, EOOD, Vratsa
- Canada (5):
  - ALTA Clinical Research Inc., Edmonton, Alberta
  - Synergy Respiratory Care, Sherwood Park, Alberta
  - Dynamic Drug Advancement, Ajax, Ontario
  - Respirology and Rheumatology Associates, Windsor, Ontario
  - C.I.C. Mauricie Inc., Trois-Rivières, Quebec
- Denmark (3):
  - Hvidovre Hospital, Hvidovre
  - Odense Universitetshospital, Odense C
  - Zealand University Hospital, Roskilde, Roskilde
- Tartu University Hospital, Lung Clinic, Tartu, Estonia
- Hungary (6):
  - Dr. Kenessey Albert Kórház-Rendelőintézet, Pulmonológiai Osztály, Balassagyarmat
  - Komlói Egészségcentrum, Bányászati Utókezelő és Éjjeli Szanatórium Egészségügyi Központ, Komló
  - Da Vinci Klinika Infer-Med Kft. Tüdőgyógyászat, Pécs
  - Szarvasi Tüdőgyógyász Kft, Szarvas
  - Csanád-Csongrád Megyei Mellkasi Betegségek Szakkórháza, Tüdőgondozó Intézet, Szeged
  - Szent Borbála Kórház, Tüdőgyógyászat, Tatabánya
- Poland (8):
  - Centrum Medyczne All-Med, Krakow
  - Małopolskie Centrum Alergologii, Krakow
  - ETG Łódź, Lodz
  - Ostrowieckie Centrum Medyczne spółka cywilna Anna Olech-Cudzik, Krzysztof Cudzik, Ostrowiec Świętokrzyski
  - Prywatny Gabinet Lekarski, Rzeszów
  - Gabinet Pulmonologii i Diagnostyki Chorób Alergicznych, Szczecin
  - Centrum Badań Klinicznych Piotr Napora Lekarze Spółka Partnerska, Wroclaw
  - "ALL-MED" Specjalistyczna Opieka Medyczna, Medyczny Instytut Badawczy, Wroclaw
- Slovakia (4):
  - Pneumologicko-ftizeologická ambulancia, Pneumomed, s.r.o, Bratislava
  - Zeleznicna nemocnica s poliklinikou, Košice
  - Ambulancia pneumologie a ftizeologie, ZAPA JJ, s.r.o., Levice
  - Univerzitna nemocnica Martin, Klinika pneumologie a ftizeologie, Martin
- Spain (4):
  - Hospital Vithas Internacional Xanit, Benalmádena, Málaga
  - Institut Catala de Serveis Medics, Girona
  - Hospital Clinico Universitario Virgen de la Victoria, Málaga
  - Hospital Clinico Universitario de Valencia, Valencia

REFERENCES:
- [Derived] Dransfield M, Marchetti N, Kalhan R, Reyner D, Dixon AL, Rheault T, Rickard KA, Anzueto A. Ensifentrine in COPD patients taking long-acting bronchodilators: A pooled post-hoc analysis of the ENHANCE-1/2 studies. Chron Respir Dis. 2025 Jan-Dec;22:14799731251314874. doi: 10.1177/14799731251314874. PMID 39854278
- [Derived] Sciurba FC, Christenson SA, Rheault T, Bengtsson T, Rickard K, Barjaktarevic IZ. Effect of Dual Phosphodiesterase 3 and 4 Inhibitor Ensifentrine on Exacerbation Rate and Risk in Patients With Moderate to Severe COPD. Chest. 2025 Feb;167(2):425-435. doi: 10.1016/j.chest.2024.07.168. Epub 2024 Aug 27. PMID 39197510
- [Derived] Mahler DA, Bhatt SP, Rheault T, Reyner D, Bengtsson T, Dixon A, Rickard K, Singh D. Effect of ensifentrine on dyspnea in patients with moderate-to-severe chronic obstructive pulmonary disease: pooled analysis of the ENHANCE trials. Expert Rev Respir Med. 2024 Aug;18(8):645-654. doi: 10.1080/17476348.2024.2389960. Epub 2024 Aug 8. PMID 39106052
- [Derived] Anzueto A, Barjaktarevic IZ, Siler TM, Rheault T, Bengtsson T, Rickard K, Sciurba F. Ensifentrine, a Novel Phosphodiesterase 3 and 4 Inhibitor for the Treatment of Chronic Obstructive Pulmonary Disease: Randomized, Double-Blind, Placebo-controlled, Multicenter Phase III Trials (the ENHANCE Trials). Am J Respir Crit Care Med. 2023 Aug 15;208(4):406-416. doi: 10.1164/rccm.202306-0944OC. PMID 37364283

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This Phase 3, randomized, double-blind, placebo-controlled study was conducted in patients with moderate to severe chronic obstructive pulmonary disease (COPD) at 130 study centers in Belgium, Bulgaria, Canada, Denmark, Estonia, Hungary, Poland, Slovakia, Spain, United States of America between 22 September 2020 and 06 July 2022. Patients were randomized in a 5:3 ratio, stratified by smoking status and background medication use, manner to receive either ensifentrine or placebo.
Pre-assignment Details: Patients were screened for eligibility before entering a 28-day run in period to ensure a stable COPD treatment regimen and to collect baseline information on symptoms and rescue medication use.
Groups:
- Ensifentrine: 3 mg twice daily via standard jet nebulizer
- Placebo: twice daily via standard jet nebulizer
Period: Overall Study
Arm/Group | Ensifentrine | Placebo
Started | 499 | 291
Received Treatment | 498 | 291
Completed | 393 | 218
Not Completed | 106 | 73
Not completed — Death | 3 | 1
Not completed — COPD exacerbation withdrawal criteria | 5 | 6
Not completed — Coronavirus disease 2019 (COVID-19) | 10 | 7
Not completed — Adverse Event | 15 | 6
Not completed — COVID-19 adverse event | 6 | 4
Not completed — Lack of Efficacy | 2 | 5
Not completed — Study terminated by sponsor | 1 | 0
Not completed — Investigator discretion | 2 | 1
Not completed — Withdrawal by Subject | 52 | 30
Not completed — Lost to Follow-up | 8 | 11
Not completed — Other | 2 | 2

BASELINE CHARACTERISTICS:
Population: All patients randomized set included all patients in the enrolled set who were randomized to study medication.
Groups:
- Total: Total of all reporting groups
Arm/Group | Ensifentrine | Placebo | Total
Number analyzed (Participants) | 499 | 291 | 790
Age, Continuous [Mean (Standard Deviation); unit: years] | 65.0 (7.38) | 65.3 (7.30) | 65.1 (7.35)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 254 | 153 | 407
  Male | 245 | 138 | 383
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  American Indian or Alaska native | 1 | 0 | 1
  Asian | 1 | 1 | 2
  Black or African American | 24 | 11 | 35
  White | 472 | 276 | 748
  Other | 1 | 3 | 4
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Hispanic or Latino | 26 | 14 | 40
  Not Hispanic or Latino | 473 | 277 | 750
Region of Enrollment [Number; unit: participants]
  Belgium | 4 | 1 | 5
  Bulgaria | 78 | 53 | 131
  Canada | 7 | 6 | 13
  Denmark | 3 | 1 | 4
  Estonia | 18 | 2 | 20
  Hungary | 32 | 20 | 52
  Poland | 38 | 20 | 58
  Slovakia | 13 | 5 | 18
  Spain | 25 | 9 | 34
  United States | 281 | 174 | 455

OUTCOME MEASURES:

1. Primary Outcome: Least Square (LS) Mean Change From Baseline in Average Forced Expiratory Volume in 1 Second (FEV1) Area Under the Curve Over 12 Hours (AUC0-12h) at Week 12
Description: Forced spirometry maneuvers including the FEV1 were used to assess pulmonary function. Average FEV1 AUC0-12h was defined as AUC over 12 hours of the FEV1, divided by 12 hours. Baseline FEV1 is the mean of the 2 measurements taken before study medication on the day of first dosing, that is, <=40 minutes pre-dose on Day 1. Spirometry assessments were performed in accordance with American Thoracic Society (ATS)/European Respiratory Society (ERS) guidelines.
Time Frame: Baseline (40 minutes before first administration on Day 1) and Week 12
Population: The modified Intent-to-Treat (mITT) population set included all patients in the randomized set who received at least 1 dose (or partial dose) of study medication, and patients were classified according to randomized treatment.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Ensifentrine | Placebo
Number analyzed (Participants) | 498 | 291
liters | 0.0480 (0.00941) | -0.0462 (0.01236)
Statistical Analysis 1: Comparison: Ensifentrine vs Placebo; Test type: Superiority; p < 0.0001, ANCOVA — The analysis of covariance (ANCOVA) model was used to model the change from baseline FEV1 to average FEV1 AUC0-12h with treatment, region, background medication strata and smoking strata as fixed effects and baseline FEV1 as covariate; LS mean difference = 0.0941, 95% CI 2-sided [0.0647 to 0.1236], Standard Error of Mean 0.01501

2. Secondary Outcome: LS Mean Change From Baseline FEV1 to Peak FEV1 at Day 1 and Weeks 6, 12 and 24
Description: Forced spirometry maneuvers including the FEV1 were used to assess pulmonary function. Peak FEV1 is the maximum value in the 4 hours after dosing. Baseline FEV1 is the mean of the 2 measurements taken before study medication on the day of first dosing, that is, <=40 minutes pre-dose on Day 1. Spirometry assessments were performed in accordance with ATS/ERS guidelines.
Time Frame: Baseline (40 minutes before first administration on Day 1), post-dose on Day 1, Weeks 6, 12, and 24
Population: The mITT population set included all patients in the randomized set who received at least 1 dose (or partial dose) of study medication, and patients were classified according to randomized treatment.
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Ensifentrine | Placebo
Number analyzed (Participants) | 498 | 291
liters
  Day 1 (Post-dose) | 0.2369 (0.00601) | 0.0801 (0.00784)
  Week 6 | 0.2158 (0.00969) | 0.0636 (0.01276)
  Week 12 | 0.1945 (0.01012) | 0.0482 (0.01349)
  Week 24 | 0.1957 (0.01099) | 0.0434 (0.01475)

3. Secondary Outcome: LS Mean Change From Baseline to the Mean Weekly Evaluating-Respiratory Symptoms (E-RS) Total Score at Weeks 6, 12 and 24
Description: The E-RS scale consists of 11 questions, with 3 sub-domains of: breathlessness, cough and sputum, and chest symptoms. The E-RS sub-domain score was calculated as the sum from the relevant questions. The E-RS total score was derived as the sum of the raw scores of the 11 items ranging from 0 to 40. Higher scores indicates severe respiratory symptoms. Scores were derived weekly as the mean over 7 days prior to the visit, using only days where data was recorded. The E-RS was collected daily by electronic diary (e-diary). Baseline is the mean over the 7 days prior to the first intake of study medication, using only days where data was recorded.
Time Frame: Baseline (average of 7 days before first administration on Day 1) and Weeks 6, 12, and 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ensifentrine | Placebo
Number analyzed (Participants) | 492 | 291
units on a scale
  Week 6 | -1.938 (0.2086) | -0.614 (0.2763)
  Week 12 | -2.051 (0.2245) | -1.161 (0.2963)
  Week 24 | -2.146 (0.2557) | -1.529 (0.3365)

4. Secondary Outcome: LS Mean Change From Baseline in the St. George's Respiratory Questionnaire (SGRQ) Total Score at Weeks 6, 12 and 24
Description: The SGRQ questionnaire consists of 17 questions, split into 2 parts. Part 1 consisted of the first 8 questions and was related to the symptoms subdomain. The remaining 9 questions were in Part 2, which were related to the activity and impacts subdomains. The total score was calculated by dividing the summed weights by the maximum possible weight for all items in the questionnaire and expressing the result as a percentage. Score ranging from 0 to 100 and higher scores indicated a worse outcome. Baseline is the score calculated on Day 1 prior to 4 hour post-dose spirometry.
Time Frame: Baseline (40 minutes before first administration on Day 1) and Weeks 6, 12, and 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ensifentrine | Placebo
Number analyzed (Participants) | 489 | 286
units on a scale
  Week 6 | -3.602 (0.5902) | -1.890 (0.7692)
  Week 12 | -4.019 (0.6171) | -2.942 (0.8168)
  Week 24 | -4.532 (0.6840) | -4.054 (0.9084)

5. Secondary Outcome: LS Mean Change From Baseline FEV1 to Morning Trough FEV1 at Weeks 6, 12 and 24
Description: Forced spirometry maneuvers including the FEV1 were used to assess pulmonary function. Morning trough FEV1 was the last value collected prior to the morning dose. Baseline FEV1 is the mean of the two measurements taken before study medication on the day of first dosing, that is, <=40 minutes pre-dose on day 1. Spirometry assessments were performed in accordance with ATS/ERS guidelines.
Time Frame: Baseline (40 minutes before first administration on Day 1) and Weeks 6, 12, and 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Ensifentrine | Placebo
Number analyzed (Participants) | 498 | 291
liters
  Week 6 | 0.0177 (0.00899) | -0.0261 (0.01181)
  Week 12 | 0.0057 (0.00957) | -0.0435 (0.01266)
  Week 24 | -0.0066 (0.01006) | -0.0318 (0.01323)

6. Secondary Outcome: LS Mean Change From Baseline in Average FEV1 Area Under the Curve Over 4 Hours (AUC0-4h) at Day 1 and Weeks 6, 12 and 24
Description: Forced spirometry maneuvers including the FEV1 were used to assess pulmonary function. Average FEV1 AUC0-4h was defined as area under the curve over 4 hours of the FEV1, divided by 4 hours. Baseline FEV1 is the mean of the 2 measurements taken before study medication on the day of first dosing, that is, <=40 minutes pre-dose on Day 1. Spirometry assessments were performed in accordance with ATS/ERS guidelines.
Time Frame: Baseline (40 minutes before first administration on Day 1), post-dose on Day 1, Weeks 6, 12, and 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Ensifentrine | Placebo
Number analyzed (Participants) | 498 | 291
liters
  Day 1 (Post-dose) | 0.1556 (0.00527) | 0.0063 (0.00686)
  Week 6 | 0.1357 (0.00932) | -0.0082 (0.01209)
  Week 12 | 0.1148 (0.00943) | -0.0209 (0.01260)
  Week 24 | 0.1148 (0.01036) | -0.0248 (0.01381)

7. Secondary Outcome: Percentage of SGRQ Responders at Weeks 6, 12 and 24
Description: The SGRQ questionnaire consists of 17 questions, split into 2 parts. Part 1 consisted of the first 8 questions and was related to the symptoms subdomain. The remaining 9 questions were in Part 2, which were related to the activity and impacts subdomains. The total score was calculated by dividing the summed weights by the maximum possible weight for all items in the questionnaire and expressing the result as a percentage. Responder was a patient with an improvement from baseline in SGRQ total score of 4 or more. Percentage of SGRQ responders are reported.
Time Frame: Weeks 6, 12 and 24
Population: as for outcome 2
Measure: Number; unit: percentage of patients
Arm/Group | Ensifentrine | Placebo
Number analyzed (Participants) | 489 | 286
percentage of patients
  Week 6 | 44.0 | 39.5
  Week 12 | 45.2 | 43.0
  Week 24 | 45.4 | 50.3

8. Secondary Outcome: LS Mean Change From Baseline to the Mean Weekly Rescue Medication Use at Weeks 6, 12 and 24
Description: Use of rescue medication (albuterol/salbutamol) per week was calculated as the LS mean use daily over 7 days. Daily rescue medication use was collected in an e-diary throughout the study. Baseline is the mean over the 7 days prior to the first intake of study medication, calculated as the sum of puffs taken, divided by number of days data has been recorded.
Time Frame: Baseline (average of 7 days before first administration on Day 1) and Weeks 6, 12, and 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: avg number of rescue medication puffs
Arm/Group | Ensifentrine | Placebo
Number analyzed (Participants) | 492 | 291
avg number of rescue medication puffs
  Week 6 | -0.530 (0.0883) | -0.191 (0.1165)
  Week 12 | -0.573 (0.0745) | -0.288 (0.0976)
  Week 24 | -0.485 (0.0871) | -0.346 (0.1143)

9. Secondary Outcome: LS Mean Transition Dyspnea Index (TDI) Questionnaire Total Score at Weeks 6, 12 and 24
Description: The TDI is a questionnaire that focused on 3 sub-domains: functional impairment, magnitude of task and magnitude of effort. Sub-domain score was calculated as the sum from the related questions. Total score was calculated as the sum of the sub-domain scores. The TDI measures the change in dyspnea severity from the baseline as measured by the baseline dyspnea index. It was rated by 7 grades ranging from -3 (major deterioration) to +3 (major improvement). Higher scores indicate better outcome. Change from baseline was assessed with the Baseline Dyspnea Index.
Time Frame: Weeks 6, 12 and 24
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: units on a scale
Arm/Group | Ensifentrine | Placebo
Number analyzed (Participants) | 484 | 286
units on a scale
  Week 6 | 1.6 (0.12) | 0.9 (0.16)
  Week 12 | 1.8 (0.13) | 1.2 (0.18)
  Week 24 | 2.2 (0.15) | 1.3 (0.20)

10. Secondary Outcome: LS Mean Change From Baseline FEV1 to Evening Trough FEV1 at Week 12
Description: Forced spirometry maneuvers including the FEV1 were used to assess pulmonary function. Evening trough FEV1 was the value collected at 12 hours post-morning dose and prior to the evening dose. Baseline FEV1 is the mean of the 2 measurements taken before study medication on the day of first dosing, that is, <=40 minutes pre-dose on day 1. Spirometry assessments were performed in accordance with ATS/ERS guidelines.
Time Frame: Baseline (40 minutes before first administration on Day 1) and Week 12
Population: as for outcome 2
Measure: Least Squares Mean (Standard Error); unit: liters
Arm/Group | Ensifentrine | Placebo
Number analyzed (Participants) | 498 | 291
liters | -0.0246 (0.01079) | -0.0783 (0.01358)

ADVERSE EVENTS:
Time Frame: Treatment-emergent adverse events (TEAEs) were collected from the first dose of study treatment up to 10 days after the final study visit at Week 24, approximately 25 weeks.
Description: The safety analysis set included all patients in the randomized set who received at least 1 dose (or partial dose) of study medication, and patients were classified according to treatment received. The TEAEs defined as adverse events that started or worsened in severity on or after the first dose of study treatment are reported.
Arm/Group | Ensifentrine | Placebo
All-Cause Mortality (participants affected / at risk) | 4/498 | 1/291
Serious Adverse Events (participants affected / at risk) | 28/498 | 17/291
Other Adverse Events (participants affected / at risk) | 68/498 | 46/291
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Ensifentrine (N=498) | Placebo (N=291)
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 10 | 5
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 0 — Acute respiratory failure secondary to these adverse events: COVID-19 pneumonia, acute diastolic congestive heart failure, and toxicity to various agents.
Bronchiectasis (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Interstitial lung disease (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 1
Pneumonia (Infections and infestations) | 2 | 4
COVID-19 pneumonia (Infections and infestations) | 2 | 2
Clostridium difficile infection (Infections and infestations) | 0 | 1
Colonic abscess (Infections and infestations) | 1 | 0
Erysipelas (Infections and infestations) | 1 | 0
Septic shock (Infections and infestations) | 0 | 1
Sinusitis (Infections and infestations) | 1 | 0
Urinary tract infection (Infections and infestations) | 1 | 0
Basal cell carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Bladder cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Laryngeal cancer stage II (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Lung neoplasm malignant (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
Oesophageal neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
Ankle fracture (Injury, poisoning and procedural complications) | 1 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1
Overdose (Injury, poisoning and procedural complications) | 1 | 0
Toxicity to various agents (Injury, poisoning and procedural complications) | 1 | 0
Acute left ventricular failure (Cardiac disorders) | 1 | 0
Atrial fibrillation (Cardiac disorders) | 1 | 0
Coronary artery disease (Cardiac disorders) | 0 | 1
Myocardial ischaemia (Cardiac disorders) | 0 | 1
Adverse drug reaction (General disorders) | 1 | 0
Chest pain (General disorders) | 1 | 0
Vertigo positional (Ear and labyrinth disorders) | 1 | 0
Hemiparesis (Nervous system disorders) | 1 | 0
Suicide attempt (Psychiatric disorders) | 1 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 1% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Ensifentrine (N=498) | Placebo (N=291)
COVID-19 (Infections and infestations) | 16 | 10
Urinary tract infection (Infections and infestations) | 7 | 5
Nasopharyngitis (Infections and infestations) | 9 | 3
Sinusitis (Infections and infestations) | 5 | 0
Dyspnea (Respiratory, thoracic and mediastinal disorders) | 3 | 4
Diarrhea (Gastrointestinal disorders) | 8 | 2
Back pain (Musculoskeletal and connective tissue disorders) | 8 | 5
Headache (Nervous system disorders) | 10 | 7
Angina pectoris (Cardiac disorders) | 1 | 4
Hypertension (Vascular disorders) | 5 | 1
Vertigo (Ear and labyrinth disorders) | 1 | 3
Tooth Abcess (Infections and infestations) | 0 | 4
Gastrooesophageal reflux disease (Gastrointestinal disorders) | 2 | 3

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes

DOCUMENTS (2):
  • Study Protocol (2021-04-30): https://cdn.clinicaltrials.gov/large-docs/57/NCT04542057/Prot_000.pdf
  • Statistical Analysis Plan (2022-07-25): https://cdn.clinicaltrials.gov/large-docs/57/NCT04542057/SAP_001.pdf